CLINICAL TRIAL: NCT00165061
Title: Phase 3 Multicenter Randomized Study Comparing Esophagectomy Against Definitive Chemoradiation for Treatment of Squamous Esophageal Cancer
Brief Title: Multi-Center Prospective Randomized Trial Comparing Standard Esophagectomy Against Chemo-Radiotherapy for Treatment of Squamous Esophageal Cancer - Early Results From the Chinese University Research Group for Esophageal Cancer (CURE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE-9362
Record Dates: First submitted 2005-09-13; First posted 2005-09-14 (Estimated); Last update posted 2005-09-14 (Estimated); Status verified 2005-09

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy; Chemoradiotherapy

INTERVENTIONS:
Procedure: Esophagectomy
Procedure: Chemoradiation

SUMMARY:
A multicenter randomized comparison of primary esophagectomy against definitive chemoradiotherapy for the treatment of squamous esophageal cancer.

DETAILED DESCRIPTION:
Cancer of the oesophagus is notorious for its grave prognosis with an overall 5-year survival rate of 10-20%. Surgical resection with curative intent remains the most effective treatment for this disease. To improve the survival, a better treatment approach is in need to manage patients with oesophageal cancer. Unfortunately, the use of preoperative adjuvant chemotherapy or adjuvant radiotherapy does not confer any survival benefit to patients with localized oesophageal cancer as proven in most randomized studies. However, the combination of chemotherapy and radiotherapy has greater clinical efficacy in achieving complete pathological regression of the tumour as well as the response rate as shown in our preliminary results. In fact, treatment of squamous oesophageal cancer by primary chemo-irradiation without surgery is now feasible.

We propose to conduct a multi-center randomized trial to evaluate the efficacy and the patients' survival by comparing primary chemo-irradiation without surgery versus standard surgical resection as the treatment for squamous oesophageal cancer. Those patients with residual cancer after primary chemo-irradiation will have salvage oesophagectomy to control the disease. Over a 3-year period, a total of 80 patients will be recruited from 4 different hospitals with 100 patients being randomized into each treatment arm. Treatment outcomes will be compared on an intention-to-treat analysis basis.

ELIGIBILITY:
Inclusion Criteria:

* mid or lower thoracic esophageal cancers that were confirmed on histology to be a squamous cell carcinoma deemed to be resectable

Exclusion Criteria:

* distant metastasis to solid visceral organs
* local invasion into trachea, descending aorta or recurrent laryngeal nerve.
* patients > 75 years
* serious premorbid condition
* poor physical status that compromised a thoracotomy
* compromised cardiac function
* creatinine clearance less than 50 ml/min were not eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2000-07

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
1.Disease free survival
2.Hospital stay
3.Morbidities
4.Recurrence of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Philip WY Chiu, MBChB, FRCSEd, Principal Investigator — Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong; Angus CW Chan, MD, Study Director — Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong
Locations (1):
- Department of Surgery, Prince of Wales Hospital, The Chinese University of Hong Kong, Hong Kong, China